CLINICAL TRIAL: NCT04572815
Title: Randomized, Placebo-Controlled, Phase II Trial Examining Ustekinumab for Prevention of Graft Vs. Host Disease After Allogeneic Hematopoietic Cell Transplantation
Brief Title: Ustekinumab for the Prevention of Acute Graft-versus-Host Disease After Unrelated Donor Hematopoietic Cell Transplant
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RG1005588; NCI-2020-02617 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10421 (Other: Fred Hutch/University of Washington Cancer Consortium); R01FD006836 (FDA)
Record Dates: First submitted 2020-09-28; First posted 2020-10-01 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Hematologic and Lymphocytic Disorder; Hematopoietic and Lymphoid System Neoplasm
MeSH Terms: conditions — Hematologic Diseases | interventions — Ustekinumab; Immunoglobulin G; Interleukin-12 Subunit p40; Disulfides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ustekinumab) (Experimental): Between 4 and 72 hours prior to start of HCT conditioning therapy, patients receive ustekinumab IV. Beginning 8 weeks after receiving IV ustekinumab, patients receive ustekinumab SC on days 50 (+/- 5 days), 100 (+/- 7 days), and 160 (+/- 7 days) post-HCT in the absence of grade III-IV acute GVHD, disease relapse or unacceptable toxicity. NOTE: HCT infusion takes place on day 0.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Biological: Ustekinumab
- Arm II (placebo) (Placebo Comparator): Between 4 and 72 hours prior to start of HCT conditioning therapy, patients receive a placebo IV. Beginning 8 weeks after IV placebo, patients receive a placebo SC on days 50 (+/- 5 days), 100 (+/- 7 days), and 160 (+/- 7 days) post-HCT in the absence of grade III-IV acute GVHD, disease relapse, or unacceptable toxicity. NOTE: HCT infusion takes place on day 0.
  Interventions: Drug: Placebo Administration; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Placebo Administration — Given IV and SC
  Arms: Arm II (placebo)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Biological: Ustekinumab — Given IV and SC
  Other Names: CNTO 1275; CNTO1275; Immunoglobulin G1, Anti-(Human Interleukin-12 Subunit beta (IL-12B, CLMF p40, NKSF2)) (Human Monoclonal CNTO 1275 gamma1-chain), Disulfide with Human Monoclonal CNTO 1275 kappa-chain, Dimer; Stelara
  Arms: Arm I (ustekinumab)

SUMMARY:
This phase II trial studies how well ustekinumab works in preventing acute graft-versus-host disease after unrelated donor hematopoietic cell transplant. Sometimes the transplanted cells from a donor can attack the body's normal tissues (called graft-versus-host disease). Giving ustekinumab after the transplant may help prevent acute graft-versus-host disease by controlling the body's immune response. Funding Source- FDA OOPD.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Between 4 and 72 hours prior to start of HCT conditioning therapy, patients receive ustekinumab intravenously (IV). Beginning 8 weeks after receiving IV ustekinumab, patients receive ustekinumab subcutaneously (SC) on days 50 (+/- 5 days), 100 (+/- 7 days), and 160 (+/- 7 days) post-HCT in the absence of grade III-IV acute GVHD, disease relapse or unacceptable toxicity. NOTE: HCT infusion takes place on day 0.

ARM II: Between 4 and 72 hours prior to start of HCT conditioning therapy, patients receive a placebo IV. Beginning 8 weeks after IV placebo, patients receive a placebo SC on days 50 (+/- 5 days), 100 (+/- 7 days), and 160 (+/- 7 days) post-HCT in the absence grade III-IV acute GVHD, of disease relapse, or unacceptable toxicity. NOTE: HCT infusion takes place on day 0.

After completion of study, patients are followed up at 6, 9, 12, 18, and 24 months post-HCT.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 70
* Signed informed consent.
* Hematologic malignancy or disorder requiring allogeneic hematopoietic cell transplantation
* Adequate vital organ function:

  1. Left ventricular ejection fraction (LVEF) ≥ 50%
  2. Forced expiratory volume in 1 second (FEV1), forced vital capacity (FVC), and diffusion capacity of the lung for carbon monoxide (DLCO) ≥ 50% of predicted values on pulmonary function tests
  3. Transaminases (aspartate aminotransferase [AST], aspartate aminotransferase [ALT]) < 3 times upper limit of normal values
  4. Creatinine clearance ≥ 50 cc/min.
* Performance status: Karnofsky Performance Status Score ≥ 70%.
* HCT donor is at least 8/8 (matched at HLA-A, -B, -C, -DRB1) matched with the recipient
* PBSC (peripheral blood mobilized stem cells) as graft source
* Fully myeloablative, reduced-toxicity ablative, or reduced-intensity conditioning regimens. If melphalan is part of the conditioning regimen, dose must be at least 75mg/m^2

Exclusion Criteria:

* Active infection not controlled with appropriate antimicrobial therapy
* Human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection
* Anti-thymocyte globulin (ATG) as part of the conditioning regimen or GVHD prophylaxis
* Pregnant or nursing women
* Subjects of childbearing age unwilling to use an effective birth control method or refrain from sexual intercourse until 15 weeks after last dose of study drug
* Non-myeloablative conditioning regimens or conditioning regimens that use less than 75mg/m^2 of melphalan
* Prior allogeneic transplant
* Non-malignant blood disorders (e.g. sickle cell disease, aplastic anemia)
* Positive screening test for tuberculosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-05-14 (Actual); Primary Completion 2025-10-27 (Actual); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Grade II-IV acute graft versus host disease (GVHD) survival | At 6 months post-hematopoietic cell transplantation (HCT)
  Will be treated as a binary outcome, and the Cochran-Mantel-Haenszel test will be used to compare the two groups based on the stratification factors.

SECONDARY OUTCOMES:
Cumulative incidence of grade II-IV and grade III-IV acute GVHD | At 100 days post-HCT
Cumulative incidence of grade II-IV and grade III-IV acute GVHD | At 6 months post-HCT
Acute GVHD organ staging, overall grading, and classification | From time of HCT, assessed up to day 100 post-HCT
  Minnesota risk criteria will be used to assess organ involvement, individual organ staging, and overall acute GVHD grade. Risk classification will be performed per MacMillan et al.
Incidence of overall chronic GVHD | From time of HCT, assessed up to 2 years post-HCT
  Will be assessed at serial study visits, and scored according to National Institutes of Health Consensus criteria.
Incidence of moderate-severe chronic GVHD | From time of HCT, assessed up to 2 years post-HCT
  Will be assessed at serial study visits, and scored according to National Institutes of Health Consensus criteria.
Incidence of post-HCT relapse | From time of HCT, assessed up to 2 years post-HCT
  Relapse is defined as hematologic relapse or any unplanned intervention (including withdrawal of immune suppression) to prevent progression of disease in patients with evidence (molecular, cytogenetic, flow cytometric, radiographic) of malignant disease. Will be compared using either the log-rank test (if no competing risks) or Gray's test (if competing risks are present). For time-to-event endpoints with competing risks, the log-rank test will also be used for exploratory purposes.
Incidence of non-relapse mortality | From time of HCT, assessed up to 2 years post-HCT
  Non-relapse mortality indicates death with primary malignancy that served as HCT indication in remission. Will be compared using either the log-rank test (if no competing risks) or Gray's test (if competing risks are present). For time-to-event endpoints with competing risks, the log-rank test will also be used for exploratory purposes.
Relapse-free survival | From time of HCT, assessed up to 2 years post-HCT
  Relapse is defined as hematologic relapse or any unplanned intervention (including withdrawal of immune suppression) to prevent progression of disease in patients with evidence (molecular, cytogenetic, flow cytometric, radiographic) of malignant disease. Will be compared using either the log-rank test (if no competing risks) or Gray's test (if competing risks are present). For time-to-event endpoints with competing risks, the log-rank test will also be used for exploratory purposes.
Overall survival | From time of HCT, assessed up to 2 years post-HCT
  Will be compared using either the log-rank test (if no competing risks) or Gray's test (if competing risks are present). For time-to-event endpoints with competing risks, the log-rank test will also be used for exploratory purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie J. Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (4):
- United States (4):
  - City of Hope Comprehensive Cancer Center,, Duarte, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/15/NCT04572815/ICF_000.pdf